CLINICAL TRIAL: NCT02155764
Title: Comparison of Octacalcium Phosphate Synthetic Bone Graft (OctoFor) and Bovine-derived Bone (Bio-Oss) for Ridge Preservation After Tooth Extraction: Open, Prospective, Non-Randomised Clinical Trial
Brief Title: Ridge Preservation With New Class of Osteoplastic Materials
Acronym: RP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Collaborators: Central Scientific Research Institute of Dentistry and Maxillo-facial Surgery, Moscow, Russia (Unknown); Bionova, Skolkovo Community, Russia (Unknown)
Responsible Party: Principal Investigator, Alex Gurin, Teaching Assistant, PhD, I.M. Sechenov First Moscow State Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11-13; 11-13 (Other: The I.M. Sechenov Moscow Medical Academy)
Record Dates: First submitted 2014-05-29; First posted 2014-06-04 (Estimated); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Tooth Extraction; Atrophy of Edentulous Alveolar Ridge
Keywords: tooth; extraction; alveolar socket; socket preservation; ridge preservation; bone graft; tricalcium phosphate; octacalcium phosphate; xenograft; bio oss

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Octacalcium phosphate (Experimental): Bone augmentation, after tooth extraction, with Octacalcium phosphate (synthetic bone graft material) in combination with resorbable collagen membrane Bio-Gide.
  Interventions: Device: Octacalcium phosphate
- Bio-Oss (Active Comparator): Bone augmentation, after tooth extraction, with Bio-Oss (bovine-derived xenograft)in combination with resorbable collagen membrane Bio-Gide
  Interventions: Device: Bio-Oss
- Tricalcium phosphate (Active Comparator): Bone augmentation, after tooth extraction, with Tricalcium phosphate (synthetic bone graft material) in combination with resorbable collagen membrane Bio-Gide.
  Interventions: Device: Tricalcium phosphate

INTERVENTIONS:
Device: Octacalcium phosphate — Bone augmentation, after tooth extraction, with Octacalcium Phosphate (synthetic bone graft material) in combination with resorbable collagen membrane Bio-Gide.
  Other Names: OctoFor
  Arms: Octacalcium phosphate
Device: Bio-Oss — Bone augmentation, after tooth extraction, with Bio-Oss (bovine-derived xenograft)in combination with resorbable collagen membrane Bio-Gide
  Arms: Bio-Oss
Device: Tricalcium phosphate — Bone augmentation, after tooth extraction, with Tricalcium Phosphate (synthetic bone graft material) in combination with resorbable collagen membrane Bio-Gide.
  Other Names: TriCafor
  Arms: Tricalcium phosphate

SUMMARY:
Return to normal life and shortening rehabilitation period of patients after surgical removal of teeth is important and urgent social problem. In this regard, higher demands for quality of care and treatment of patients, which requires the development of new approaches to the treatment of patients, the introduction of new technologies and the associated development of new materials . Serious problem of contemporary oral and maxillo-facial surgery and dentistry is augmentation of bone defects generated during the surgical treatment of diseases and injuries of the bones. The results of surgical repair of bone defects are more dependent on the course of the process of reparative osteogenesis. Long-term periods of clinical studies indicate that reparative osteogenesis in posttraumatic bone defects is slow - months and years, and in some cases no bone defects filled with bone tissue.

This project aims at addressing the preservation of bone volume in humans after tooth extraction using biomaterials with optimum performance. The practical significance of the project is to establish an effective tissue response and, thus, possible subsequent quality installation of dental implants. The proposed solution is based on the scientific development of the operative techniques, and a comparative analysis of several classes of biomaterials (xenogenic and synthetic analogs), including the use of biological precursors of bone apatite mineralization having osteoinductive (stimulating) properties.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have voluntarily signed the informed consent
* Males and females, 18 years to 75 years of age
* Patient needs single tooth extraction in mandibular or maxillary incisor or pre-molar region and would benefit from prosthetic reconstruction with a dental implant
* Patients must be committed to the study and must sign informed consent
* Patient in good general health as documented by self assessment

Exclusion Criteria:

Systemic exclusion criteria:

* Patient who has any known diseases (not including controlled diabetes mellitus), infections or recent surgical procedures within 30 days of study initiation
* Female patient who are pregnant or lactating or of child bearing potential not using acceptable methods of birth control (hormonal, barriers or abstinence
* Patient who are on chronic treatment (i.e., two weeks or more) with any medication known to affect oral status (e.g., phenytoin, dihydropyridine calcium antagonists, cyclosporine, and non-steroidal anti-inflammatory drugs) within one month of baseline visit
* Patient who knowingly has HIV or Hepatitis
* Alcoholism or chronically drug abuse causing systemic compromisation
* Patient who is a heavy smoker (>10/cigarettes per day).

Local exclusion criteria

* Uncontrolled or untreated periodontal disease
* Patient who has a full mouth plaque level >30 % at the enrolment visit
* History of local radiation therapy
* Presence of oral lesions (such as ulceration, malignancy)
* Persistent intraoral infection
* Patients presenting clinical and radiological signs and symptoms of maxillary sinus disease
* Patient presents an acute endodontic lesion in the test tooth or in the neighbouring areas to the experimental procedure (sites with presence of an asymptomatic chronic lesion are eligible)

Ages: 17 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
The changes of bone level between baseline and 3 months post-extraction at the time of implantation | baseline and 3 months post-extraction
  A prefabricated stent will be used as an anchor point. After tooth extraction size of dehiscence of buccal bone from anchor point to the alveolar crest will be measured (baseline). Socket will be filled with biomaterial. After 3 months of healing at the time of implant placement the same stent will be used as an anchor point to measure size of dehiscence after socket preservation.

SECONDARY OUTCOMES:
Percent new vital bone formation | 3 month
  Bone core biopsy will be evaluated histologically for percent new vital bone formation at the time of implantation

OTHER OUTCOMES:
Percent residual graft material and percent connective tissue | 3 month
  Bone core biopsy will be evaluated histologically for percent residual bone graft material and percent connective tissue

CONTACTS AND LOCATIONS:
Overall Officials: Anatoly Kulakov, Prof, Study Director — Central Scientific Research Institute of Dentistry and Maxillo-facial Surgery
Locations (1):
- Cental Scientific Research Institute of Dentistry and Maxillo-facial Surgery, Moscow, RU, Russia

REFERENCES:
- [Background] Gurin AN, Komlev VS, Fadeeva IV, Petrakiva NV, Varda NS. [A comparative study of bone regeneration potency of alfa and beta-tricalcium phosphate bone substitute materials]. Stomatologiia (Mosk). 2012;91(6):16-21. Russian. PMID 23268211
- [Background] Gurin AN, Komlev VS, Fadeeva IV, Barinov SM. [Calcium phosphate bone cements. Application in oral and maxillofacial surgery]. Stomatologiia (Mosk). 2011;90(5):64-72. No abstract available. Russian. PMID 22332385
- [Background] Gurin AN, Komlev VS, Fadeeva IV, Barinov SM. [Octacalcium phosphate--precursor of biomineralization, novel bone scaffold]. Stomatologiia (Mosk). 2010;89(4):57-64. Russian. PMID 21186653